CLINICAL TRIAL: NCT04720859
Title: Canagliflozin: a New Therapeutic Option in Patients That Present Postprandial Hyperinsulinemic Hypoglycemia After Roux-en-Y-gastric By-pass
Brief Title: Canagliflozin in Postprandial Hyperinsulinemic Hypoglycemia (CANA-PHH-RYGB)
Acronym: CANA-PHH-RYGB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Principal Investigator, Andreea Ciudin, Associated Professor, PhD, MD, Head of the Morbid Obesity Unit, Hospital Universitari Vall d'Hebron Research Institute
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PR(AG)84/2018
Record Dates: First submitted 2021-01-19; First posted 2021-01-22 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Postprandial Hypoglycemia
MeSH Terms: conditions — Hypoglycemia | interventions — Canagliflozin; Tablets

STUDY DESIGN:
Intervention Model Description: Intervention arm in patients that present postprandial hypoglycemia following gastric by-pass and a control group of healthy subjects without intervention.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with PHH following Roux-en-Y-gastric bypass (cases) (Experimental): Patients diagnosed with PHH following Roux-en-Y-gastric bypass.
  Interventions: Drug: Canagliflozin 300 MG Oral Tablet
- Healthy individuals (controls) (No Intervention): Healthy normoweight individuals, matched by age and gender with the cases.

INTERVENTIONS:
Drug: Canagliflozin 300 MG Oral Tablet — Patients diagnosed with PHH following bariatric surgery by 100g glucose OGTT were prescribed 300mg canagliflozin during two weeks. 100g glucose OGTT response was evaluated after canagliflozin treatment.
  Arms: Patients with PHH following Roux-en-Y-gastric bypass (cases)

SUMMARY:
Roux-en-Y gastric bypass (RYGB) is the most common surgical procedure for morbid obesity. However, it can present serious late complications, like postprandial hyperinsulinemic hypoglycemia (PHH). Recent data suggested an increase in intestinal SGLT1 after RYGB. However, there are no data on the inhibition of SLGT1 to prevent PHH in patients with prior RYBG.

Objectives: To evaluate in patients that present PHH after RYGB: a) the effect of canagliflozin 300mg on the response to 100g glucose overload (OGTT); b) the pancreatic response after intra-arterial calcium stimulation.

Material and methods: Prospective pilot study, including patients with PHH after RYGB, matched by age and gender with healthy controls. Basal OGTT and after 2-weeks of daily 300mg of canagliflozin will be performed. In addition, venous sampling after intra-arterial calcium stimulation of the pancreas will be performed.

DETAILED DESCRIPTION:
A prospective opened, placebo uncontrolled, pilot interventional study is performed at the Morbid Obesity Unit of the Vall Hebron University Hospital, including patients that have previously undergone RYGB at our site and were diagnosed with PHH. The control group comprises of healthy normoweight persons matched by age, most of them family members of patients included in the study. The OGTT is performed as follows: a solution of 100g glucose was administered at 8am after 10 hours of fasting. Plasma glucose and serum insulin are measured at minute -5, +30, +60, +120, +180 after the ingestion of the glucose solution. A first OGTT is performed in basal conditions. The control group only will perform the basal OGTT. A value of plasma glucose below 50mg/dl at 60-180 minutes after the administration of the glucose solution is considered positive for PHH. The patients that additionally present a value of plasma glucose>200mg/dl during the OGTT will be selected for continuing in the study and will be prescribed canagliflozin 300mg orally daily, during 2 weeks. After 2 weeks of canagliflozin treatment, a new OGTT will be performed and, in the patients that sign the additional inform consent, the pancreatic catheterism will be realized.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with PHH following Roux-en-Y-gastric by-pass, by means of 100g Glucose OGTT. Plasma glucose <50mg/dl.
* Patients that during any time of the OGTT present at least one value of plasma glucose >200mg/dl, besides hypoglycemia

Exclusion Criteria:

* Patients unwilling to take canagliflozin 300mg
* Patients that present with PHH following other bariatric surgery techniques

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-01-05 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
response to OGTT in basal conditions and after treatment with canagliflozin 300 mg in patients with PHH after RYGB | Baseline to 180 minutes
  The OGTTis performed as follows: a solution of 100g glucose is administered at 8am after 10 hours of fasting. Plasma glucose and serum insulin were measured at minute -5, +30, +60, +120, +180 after the ingestion of the glucose solution. A first OGTT was performed in basal conditions. The control group only performed the basal OGTT. A value of plasma glucose below 50mg/dl at 60-180 minutes after the administration of the glucose solution is considered positive for PHH. The patients that additionally presented a value of plasma glucose>200mg/dl during the OGTT were selected for continuing in the study and were prescribed canagliflozin 300mg orally daily, during two weeks, and 100g glucose OGTT was repeated.

SECONDARY OUTCOMES:
Presence of nesidioblastosis | 30 minutes
  By evaluating pancreatic response to intra-arterial calcium stimulation. The right femoral artery is catheterized with another 4.1 Fr, followed by standard pancreatic arteriography, with selective injections of nonionic contrast agent into the superior mesenteric artery, gastroduodenal artery, splenic artery and common hepatic artery. Following each selective arteriogram, 10% calcium gluconate solution is diluted with normal saline into a 5 mL bolus and injected into the selective artery at a dose of 0.010-0.025 mEq Ca2+/kg. A >2-fold gradient in insulin concentration at 30, 60, 90 or 120 seconds after the arterial calcium injection and baseline in any of the superior mesenteric artery, gastroduodenal artery, splenic artery and common hepatic artery was defined as a positive response for endogenous hyperinsulinism.

CONTACTS AND LOCATIONS:
Overall Officials: Andreea Ciudin, Prof., Principal Investigator — Vall Hebron University Hospital
Locations (1):
- Andreea Ciudin, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No